CLINICAL TRIAL: NCT06354699
Title: POPSICLE (Postoperative Pain Study in Children - a Longitudinal Evaluation)
Brief Title: A Longitudinal Study Looking at the Prevalence, Risk Factors & Consequences of Persistent Post-surgical Pain in Children
Acronym: POPSICLE
Status: Recruiting | Type: Observational
Sponsor: Telethon Kids Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RGS0000003993
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Post-operative pain; Paediatric surgery
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group Elective: Patient is undergoing a surgical procedure for circumcision, hypospadias, orchidopexy or laparoscopic appendicectomy.
- Group Emergency: Patient is undergoing a surgical procedure for laparoscopic appendicectomy or scrotal exploration.

SUMMARY:
The purpose of this study is to investigate the prevalence, risk factors and consequences of chronic post-surgical pain in children aged 0-16 years through a number of questionnaires completed at various timepoints, from before surgery up to 1 year post surgery.

DETAILED DESCRIPTION:
The POPSICLE study is a multi-centre, international research study that will investigate the prevalence, risk factors and consequences of chronic post-surgical pain (CPSP) in children 0-16 years undergoing the following common paediatric surgeries: laparoscopic appendicectomy, scrotal exploration, orchidopexy, hypospadias repair and circumcisions. CPSP as well as risk factors and their association with chronic pain, including parent and child anxiety, pre-existing pain, peri-operative pain experience and acute post-operative management, will be assessed through a series of longitudinal questionnaires at 6 timepoints from pre-surgery to 10-12 months post-surgery. Baseline measures will be completed pre-operatively and post-surgery measures of pain and function will be undertaken at Day 2, 3-4 weeks, 3-4 months and 10-12 months post-operatively.

Chronic pain has a significant effect on children's quality of life, negatively impacting their physical, emotional and social health as well as schooling. Additionally, adolescent chronic pain is associated with higher rates of depression, anxiety, feeling of helplessness and lack of autonomy compared to healthy children. Therefore, evidence-based knowledge from this research will inform perioperative practice minimising the risk of a child going on to develop chronic post-surgical pain. This will benefit the child, their family and the healthcare system by aiding in the formulation of practice guidelines to follow high risk children more closely to treat any potential persistent pain earlier to avoid the development of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

The patient is undergoing a surgical procedure in either group elective (circumcision, hypospadias, orchidopexy, laparoscopic appendicectomy) or group emergency (laparoscopic appendicectomy, scrotal exploration)

Exclusion Criteria:

The parent and child have inadequate English language skills to understand the questionnaires

Children with significant/severe developmental or cognitive delay based on a formal diagnosis.

Families that are unable to complete the long-term follow up surveys.

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The participants will be the parents/legal guardians of children and the children themselves, aged 0-16 years old, undergoing planned or non-elective urgent surgical procedures.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
The prevalence of chronic post-surgical pain after 10- 12 months. | 12 months
  the prevalence of chronic post-surgical pain in paediatric patients after 10- 12 months.

SECONDARY OUTCOMES:
Identifying potential risk factors for chronic post-surgical pain | 12 months
  Identify potential biopsychosocial risk factors contributing or maintaining chronic post-surgical pain including parent and child anxiety, pre-existing and perioperative pain experience, acute postoperative management, surgical factors and to assess impacts on function one-year post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Britta P von Ungern-Sternberg, Principal Investigator — Telethon Kids Institute
Locations (16):
- United States (7):
  - University of California, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital of Michigan, Detroit, Michigan
  - Atrium Health-Wake Forest Baptist, Winston-Salem, North Carolina
  - Children's Medical Center (Dallas), Dallas, Texas
  - Texas childrens hospital, Houston, Texas
- Australia (6):
  - Townsville University hospital, Douglas, Queensland
  - Fiona Stanley Hospital, Perth, Western Australia
  - Telethon Kids Institute, Perth, Western Australia
  - Flinders Medical Centre, Adelaide
  - Women 's and Children's Hospital, Adelaide
  - Royal Darwin Hospital, Tiwi
- Canada (2):
  - Hospital for Sick Children, Toronto
  - British Columbia Children's Hospital, Vancouver
- Wellington Regional Hospital, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided